CLINICAL TRIAL: NCT06591689
Title: Investigation of the Relationship Between Communication Function and Gross Motor Function in Patients With Quadriparetic Cerebral Palsy
Brief Title: Relationship Between Communication and Gross Motor Function in Quadriparetic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Ali Demir, Physiotherapist, Acıbadem Atunizade Hospital
Other Study IDs: Ali Demir
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy, Spastic Quadriplegic; Communication Disorder, Childhood; Gross Motor Delay
MeSH Terms: conditions — Cerebral Palsy; Communication Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of Cases with Quadriparetic Cerebral Palsy — 20 quadriparetic cerebral palsy cases were evaluated with the Communication Function Classification System (CFCS), Pediatric Functional Independence Scale (WeeFIM) and Gross Motor Function Measure-88 (GMFM-88).

SUMMARY:
Communication problems are frequently encountered in quadriparetic cerebral palsy. Additionally, motor impairments often accompany this condition. Communication problems can also reduce the benefits gained from treatments, which in turn negatively affects individuals functional independence as motor impairments persist. In this study, the researchers aimed to examine the relationship between communication function, gross motor function and functional independence level.

DETAILED DESCRIPTION:
This study is an observational study conducted with data obtained from assessment scales and does not involve any treatment. The target population of the study consists of individuals diagnosed with quadriparetic cerebral palsy (QCP). Individuals with QCP aged 0-17 years were included in the study. Detailed medical histories were taken from the participants, and they were evaluated using the Communication Function Classification System (CFCS), the Pediatric Functional Independence Measure (WeeFIM), and the Gross Motor Function Measure-88 (GMFM-88). The aim of this study is to examine the effect of communication function on gross motor function and independence.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 0-17,
* Diagnosed with quadriparetic cerebral palsy,
* Participants and parents willing to participate in the study voluntarily.

Exclusion Criteria:

* Having different types of cerebral palsy such as dyskinetic, ataxic and mixed type,
* Having spastic diparetic or hemiparetic type cerebral palsy,
* Having any history of surgery on the musculoskeletal system,
* Having received Botulinum Toxin injections in the last 6 months

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Twenty quadriparetic cerebral palsy individuals between the ages of 0-17 were included in the study.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Communication Function Classification System (CFCS) | 1 month
  The communication functions of patients were evaluated using the "Communication Function Classification System (CFCS)." CFCS assesses the daily communication performance of individuals with cerebral palsy (CP) across five levels. It evaluates all methods that affect communication performance, such as speech, facial expressions, gestures, eye contact, facial cues, and the use of augmentative and alternative communication methods. In CFCS, Level I indicates a better condition, while Level V represents more impaired situations.
The Pediatric Functional Independence Measure (WeeFIM) | 1 month
  The Pediatric Functional Independence Measure (WeeFIM) is a useful, brief, and comprehensive assessment method for identifying the functional limitations of children with developmental disorders. It consists of 18 items under the categories of self-care, sphincter control, transfers, mobility, communication, and social interaction. Each item is scored between 1 and 7. A child receives a score of 1 when performing an item with full assistance, and a score of 7 when completing it independently, safely, and in a timely manner. Afterwards, all scores are summed to calculate a percentage of independence. The WeeFIM assessments were carried out by physiotherapists based on information obtained from families. High scores on this scale indicate a high level of independence.
The Gross Motor Function Measure-88 (GMFM-88) | 1 month
  The Gross Motor Function Measure-88 (GMFM-88) was used to determine the functional performance of children. GMFM-88 is a standardized, validated observational scale, and it is mandatory to use the user manual for scoring each item. GMFM-88 evaluates five domains: lying and rolling, sitting, crawling and kneeling, standing, and walking. Each section is assessed individually, and a percentage score is calculated. The total score is obtained by averaging the percentage scores of the five sections. The items in the sections are scored as 0, 1, 2, or 3. The GMFM-88 scores were calculated by physiotherapists in strict adherence to the user manual. Total GMFM-88 score is evaluated out of 100, and higher scores indicate good gross motor development.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.